# A 2-arm, open label, prefatory study to explore changes in nasal mucociliary clearance between smokers and never smokers and to standardize nasal scraping procedure

#### STATISTICAL ANALYSIS PLAN

Version No. 1

24 February 2017

Prepared by:

Requested by:

**INFLAMAX** Research Inc



USA

#### **TITLE PAGE**

**Study title:** A 2-arm, open label, prefatory study to explore changes in

nasal mucociliary clearance between smokers and never smokers and to standardize nasal scraping procedure.

Study code: 15-LE-001-RD

**Study type:** Exploratory study

Study drug:Not applicableTherapeutical area:Not applicable

Sponsor: INFLAMAX Research Inc

USA

**Version no., date:** Version No. 1, 24 February 2017

Statistical report

performed by:

#### **SIGNATURE PAGE**

**STUDY TITLE:** A 2-arm, open label, prefatory study to explore changes in nasal mucociliary clearance between smokers and never smokers and to standardize nasal scraping procedure.

**PROTOCOL VERSION:** Final 1.0

PROTOCOL DATE: 08-Dec-2016

#### **SAP PREPARED BY:**

dd/mmm/yyyy

dd/mmm/yyyy

dd/mmm/yyyy

Senior Biostatistician

**SAP REVIEWED BY:** 

Senior Biostatistician

**SAP APPROVED BY:** 

Project Manager

Inflamax Research

#### **TABLE OF CONTENTS**

| T | TLE P | AGE | 2 | |
|---|--------|------|--------------------------------------------|----|
| S | IGNAT | URE | PAGE3 | |
| T | ABLE ( | OF C | ONTENTS4 | |
| T | ABLE ( | OF T | ABLES5 | |
| T | ABLE ( | OF F | IGURES6 | |
| T | ABLE ( | OF L | ISTINGS6 | |
| 1 | INT | ROD | UCTION7 | |
| 2 | STU | JDY | OBJECTIVES AND ENDPOINT7 | |
| | 2.1 | Prir | nary objectives and endpoints | 7 |
| | 2.2 | Sec | condary objectives and endpoints | 7 |
| 3 | STU | JDY | DESIGN8 | |
| 4 | STU | JDY | POPULATION9 | |
| | 4.1 | Incl | usion criteria | 9 |
| | 4.2 | Exc | clusion criteria | 9 |
| 5 | STA | ATIS | FICAL METHODS11 | |
| | 5.1 | Sar | mple size | 11 |
| | 5.2 | Sta | tistical software | 11 |
| | 5.3 | Ana | alysis datasets | 12 |
| | 5.3. | .1 | Full Analysis Set (FAS) | 12 |
| | 5.3. | .2 | Per Protocol (PP) Population | 12 |
| | 5.3. | .3 | Safety Population | 12 |
| | 5.4 | Stu | dy hypothesis | 12 |
| | 5.5 | Sta | tistical analysis | 12 |
| | 5.5. | .1 | Subjects' disposition | 12 |
| | 5.5. | .2 | Demographic and other clinical assessments | 12 |
| | 5.5. | | Primary analysis | 13 |
| | 5.5. | .4 | Secondary analysis | 13 |
| | 5.6 | | sing values | 14 |
| 6 | | | CATIONS TO THE STUDY PROTOCOL14 | |
| 7 | | | DIX 1: DERIVED VARIABLES15 | |
| 8 | API | PENI | DIX 2: TABLES AND FIGURES16 | |
| 9 | ΔΡΙ | PFNI | DIX 2: LISTINGS 42 | |

#### **TABLE OF TABLES**

| Table A 1 – Subjects' disposition | 16 |
|---|---|
| Table A 2 – Demographic and anthropometric characteristics at visit 1 – FAS population | 17 |
| Table A 3 – Demographic and anthropometric characteristics at visit 1 – PP population | 18 |
| Table A 4 – Saccharin transit time – FAS population | 19 |
| Table A 5 – Saccharin transit time – PP population | 20 |
| Table A 6 – Plasma nicotine sample at Visit 3 – FAS population | 21 |
| Table A 7 – Plasma nicotine sample at Visit 3 – PP population | 22 |
| Table A 8 – Plasma nicotine sample versus STT | 23 |
| Table A 9 – Nasal scraping at visit 3 – FAS population | 28 |
| Table A 10 – Vital signs – Safety population | 29 |
| Table A 11 – Overall summary of adverse events – Safety population | 30 |
| Table A 12 – Adverse events – Safety population | 31 |
| Table A 13 – Hematology – Safety population | 32 |
| Table A 14 – Clinical chemistry – Safety population | 35 |
| Table A 15 – Urine – Safety population | 39 |
| Table A 16 – Serology at visit 1 – Safety population | 41 |

#### **TABLE OF FIGURES**

| Figure A 1 – Plasma nicotine levels versus STT by smokers and never smokers, at T0 – FAS | |
|---|---|
| population | 24 |
| Figure A 2 – Plasma nicotine levels versus STT by smokers and never smokers, at T4 – FAS | |
| population | 25 |
| Figure A 3 – Plasma nicotine levels versus STT by smokers and never smokers, at T8 – FAS | |
| population | 26 |
| Figure A 4 – Plasma nicotine levels versus STT by smokers and never smokers, at T12 – FAS | |
| population | 27 |
| TABLE OF LISTINGS | |
| Listing 1 – Subjects' disposition | 42 |
| Listing 2 – Protocol deviations | 43 |
| Listing 3 – Demographic and anthropometric characteristics at visit 1 | 44 |
| Listing 4 – Smoking history | 45 |
| Listing 5 – Medical history | 47 |
| Listing 6 – Prior and concomitant medication | 48 |
| Listing 7 – Exhaled Carbon Monoxide | 49 |
| Listing 8 – Drug/alcohol test | 50 |
| Listing 9 – Skin prick test | 51 |
| Listing 10 – Tobacco consumption | 52 |
| Listing 11 – Saccharin transit time test | 53 |
| Listing 12 – Vital signs | 54 |
| Listing 13 – Adverse events | 55 |
| Listing 14 – Serious adverse events | 56 |
| Listing 15 – Labs (hematology, chemistry and urine analysis) | 57 |

#### 1 INTRODUCTION

This Statistical Analysis Plan (SAP) was written in accordance with Eurotrials' Standard Operating Procedures (SOP) ST.CO.01-01 for Biostatistics and intends to provide guidelines from which the analysis will proceed, create a common and clear understanding of the planned analysis by all involved, clarify issues which was not clarified in the protocol, expand statistical section of the protocol, provide basis for the statistical section of the statistical report and reduce the opportunity for bias by prospectively defining analysis. This SAP was prepared by the biostatistician who will be further responsible (if possible) for the statistical analysis of the study data.

This SAP, in particular table shells and examples of figures/graphs, was reviewed and approved by the Sponsor's Representative previously to database locking and performance of the statistical analysis.

Any changes to the planned statistical methodology/definitions described on this SAP during the statistical analysis of the study data will be documented in the Statistical Report.

This document was written in accordance with the information contained in the Study Protocol 15-LE-001-RD, Version Final 1.0 of 08-Dec-2016 and eCRF version Final V1.0 of 12Jan2017.

#### 2 STUDY OBJECTIVES AND ENDPOINT

#### 2.1 Primary objectives and endpoints

The primary objectives of this study are:

- 1. To evaluate the NMC over the course of 12 hours following single use of cigarette in smokers.
- · STT value as assessed by STT test at each time point.
- 2. To compare NMC over the course of 12 hours in smokers following single use of cigarette relative to never smokers.
- · STT value as assessed by STT test at each time point.
- 3. To examine the relationship between plasma nicotine levels and STT value in smokers and never smokers.
- STT value as assed by the STT test and plasma nicotine levels at each time point.

#### 2.2 Secondary objectives and endpoints

The secondary objectives of this study are:

- 1. To standardize nasal scraping procedure using two methods.
- Collection of nasal epithelium for further histology.
- Evaluation of RNA quality and quantity.

- 2. To monitor the safety during the study.
- · Vital signs.
- Adverse events (AE).
- · Nasal and throat exam.
- Hematology, clinical chemistry and urine analysis.
- Brief physical examination.
- · Concomitant medications.

#### 3 STUDY DESIGN

This will be a single-center study in which 14 healthy adult male study participants, consisting of 7 cigarette smokers and 7 never smokers as a control group, will be enrolled. Study participants will not be replaced after being enrolled.

This study will have three visits on three separate days as described in Figure 1.



Figure 1 – Study flow chart

#### 4 STUDY POPULATION

#### 4.1 Inclusion criteria

- 1. Informed of the nature of the study and have agreed to and are able to read, review, and sign the informed consent form (ICF) prior to Screening. The subject must be willing to comply with the study procedures described in the informed consent. The informed consent document will be written in English, therefore the volunteer must have the ability to read and communicate in English.
- 2. Male subject aged ≥25 to ≤40 years old.
- 3. BMI between 18.0 kg/m<sup>2</sup> to 32.0 kg/m<sup>2</sup>, inclusive.
- 4. Judged by the Principal Investigator or designee to be in good health as documented by the medical history, physical examination, vital sign assessments, clinical laboratory assessments, and by general observations.
- 5. Belong to one of the following two groups:
  - a. Non-menthol cigarette smoker (meets all of the following criteria at Visit 1 and at Visit 2):
    - i. A positive urine cotinine test (≥200 ng/mL).
    - ii. Smoked at least 20 cigarettes per day for at least the past 5 years.
    - iii. eCO levels >10 parts per million (ppm).
    - iv. No plans to guit smoking in the next 3 months.
  - b. Never smoker (meets all of the following criteria at Visit 1 and at Visit 2):
    - i. Subject who has smoked less than 100 cigarettes throughout their lifetime and no cigarettes in the past 3 years.
    - ii. A negative urine cotinine test (<200 ng/mL).
    - iii. eCO levels ≤ 5 ppm.
- 6. Completed the Screening process within 30 days prior to Visit 2.
- 7. Availability for the entire study period and willingness to comply with study procedures, including smoking interruptions, as evidenced by a signed ICF and at Visit 2.

#### 4.2 Exclusion criteria

- 1. As per the Principal Investigator or designee's judgment, the subject cannot participate in the study for any reason (e.g., medical, psychiatric, and/or social reason).
- 2. Subject is legally incompetent, or physically or mentally incapable of giving consent (e.g., emergency situation, under guardianship, prisoners, or subjects who are involuntarily incarcerated).
- 3. Presence of confounding allergies including allergic rhinitis and non-allergic rhinitis during the course of the study based on medical history and SPT.
- 4. Clinical significant abnormality on their nasal and throat exam, at the discretion of the Principal Investigator or designee at Visit 1 and/or at Visit 2.
- 5. Cigarette smoker who smoke/use any tobacco or nicotine products (other than CC), such as cigars, pipe, menthol cigarettes or electronic cigarettes in the previous 3 months, as self-reported at Visit 1 or Visit 2.
- 6. Never smoker who smoke/use any tobacco or nicotine products, such as cigars, pipe, menthol cigarettes or electronic cigarettes in the previous 3 years, as self-reported at Visit 1 or Visit 2.

- 7. Cigarette smokers who state they will be unable to abstain from smoking for up to 24 hours.
- 8. Inability to taste sweet within 60 minutes in the STT test.
- 9. Subjects who routinely use or who have used in the previous 4 weeks nasal sprays, inhalers or other nasal products, such as nasal irrigation (for example, Neti Pot) prior to Visit 1 and/or Visit 2.
- 10. Subjects who have taken any of the following medication without the indicated minimum washout period:

| Prohibited Medication | Restriction period<br>(with Principal Investigator<br>or designee discretion) |
|---|---|
| Short-acting antihistamines including intranasal antihistamines | 3 days before Visit 1 until<br>Visit 2 |
| Long-acting antihistamines (i.e. Loratadine, Desloratadine) | 7 days before Visit 1 until<br>Visit 2 |
| Over-the-counter cough and cold preparations or sleep aids<br>containing antihistamines | 3 days before Visit 1 until<br>Visit 2 |
| Leukotriene inhibitors | 14 days before Visit 1 until<br>Visit 2 |
| Oral or intra-articular steroid | 30 days before Visit 1 until<br>Visit 2 |
| Intranasal and inhaled corticosteroids | 14 days before Visit 1 until<br>Visit 2 |
| Use of monoamine oxidase inhibitors | 14 days before Visit 1 until<br>Visit 2 |
| Decongestants | 48 hours before Visit 1until<br>Visit 2 |
| Cromolyn products | 14 days before Visit 1 until<br>Visit 2 |
| Beta-adrenergic blockers (i.e. Acebutolol, Atenolol, etc.) | 14 days before Visit 1 until<br>Visit 2 |
| Anticholinergies | 7 days before Visit 1 until<br>Visit 2 |
| Herbal or natural product remedies for allergy symptoms | On the day of Visit 1 until<br>Visit 2 |
| Short-Acting Beta Agonists | 6 hours prior to spirometry<br>(except as per protocol before<br>spirometry) |
| Long-Acting Beta Agonists | 3 days before Visit 1 until<br>Visit 2 |
| Phosphodiesterase 5 inhibitors (i.e. Sildenafil, Vardenafil,<br>Tadalafil) | 7 days before Visit 1 until<br>Visit 2 |
| Amiloride | 3 days before Visit 1 until<br>Visit 2 |
| Macrolide antibiotics | 7 days before Visit 1 until<br>Visit 2 |
| Guaifenesin | 3 days before Visit 1 until<br>Visit 2 |
| Mucolytic agents | 14 days before Visit 1 until<br>Visit 2 |
| Topical menthol products | 14 days before Visit 1 until<br>Visit 2 |
| Topical nasal medication | 4 weeks before Visit 1 until<br>Visit 2 |
| Topical ocular medication | 4 weeks before Visit 1 until<br>Visit 2 |
| Any other medication at the Principal Investigator or designee's discretion that might interfere with the endpoints or procedures. | |

Table 1 – Prohibited medication.

- 11. Subjects with evidence of COPD, Global Initiative for Chronic Obstructive Lung Disease (GOLD) stage I or greater, and a forced expiratory volume 1 / the forced vital capacity ratio (FEV1/FVC ratio) <0.7.
- 12. Any condition the Principal Investigator or designee has cause to believe would interfere with the procedures for upper or lower airway function. This could include, but is not limited to, nasal/septum deviations, or nasal polyps or nasal allergies which will be identified by the Principal Investigator or designee.
- 13. Upper or lower respiratory diseases in the 4 weeks prior to Visit 2.
- 14. History of nasal or sinus surgery in the 5 years prior to Visit 2.
- 15. As per the Principal Investigator or designee's judgment, the subject has medical conditions which require or will require in the course of the study, a medical intervention (e.g., start of treatment, surgery, hospitalization) which may interfere with the study participation and/or study results.
- 16. The subject has a positive alcohol test and/or a history of alcohol abuse that could interfere with the subject's participation in study at Visit 1 or Visit 2.
- 17. Positive urine drug screen at Visit 1 or Visit 2.
- 18. The subject has positive serology test for human immunodeficiency virus (HIV)1/2, Hepatitis B or Hepatitis C.
- 19. Subject has donated or been in receipt of whole blood or blood products within 3 months prior to Visit 1.
- 20. Subject is a current or former employee of the tobacco industry or of their first-degree relatives (spouse, legal patner, parent, sibling, and child).
- 21. Subject is an employee of the investigational site or any other parties involved in the study or of their first-degree relatives (spouse, legal patner, parent, sibling, and child).
- 22. Subject has been in receipt of last dose from another clinical study within 3 months prior to Visit 1.
- 23. Subject has been previously screened in this study.

#### 5 STATISTICAL METHODS

#### 5.1 Sample size

This is an exploratory study. This study will include 14 study participants: 7 cigarette smokers and 7 never smokers. No formal powering has occurred. However, with an expected standard deviation of 2.5 minutes, a difference in STT of 3.75 minutes can be detected.

#### 5.2 Statistical software

The statistical analyses will be conducted through the software SAS® (version 9.4, SAS Institute Inc, Cary).

#### 5.3 Analysis datasets

#### 5.3.1 Full Analysis Set (FAS)

All study participants who have at least one evaluable STT test at Visit 3 will be included in FAS population.

#### 5.3.2 Per Protocol (PP) Population

All study participants in Full Analysis Set who have no major protocol deviation will be included in the PP population.

#### 5.3.3 Safety Population

All enrolled subjects will be included in safety population.

#### 5.4 Study hypothesis

There are no statistical hypotheses to be tested for the primary analysis.

#### 5.5 Statistical analysis

All quantitative variables will be summarized through descriptive statistics namely mean, median, standard deviation, quartiles (Q1 and Q3) and minimum and maximum values. Qualitative variables will be summarized through number (n) and frequency distribution (%).

All descriptive analyses will be performed by smoker and never smoker group.

Statistical tests will be two-tailed considering a significance level of 5%.

#### 5.5.1 Subjects' disposition

The number of subjects included in this study will be described in this section. The number (n) and frequency distribution (%) of subjects who completed the study, subjects who discontinued the study and distribution for each study dataset will be also summarized by total, smoker and never smoker groups.

Subjects' disposition will be presented as described in **Table A 1** and listed in **Listing 1**. Protocol deviations will be listed by subject in **Listing 2**.

#### 5.5.2 Demographic and other clinical assessments

Demographics at visit 1 will be summarized by total number of observations (n), namely mean, median, standard deviation, quartiles (Q1 and Q3) and minimum and maximum values for continuous variables, and total number of observations, number (n) and frequency distribution (%) for categorical variables.

Demographics and other assessments will be presented for FAS and PP dataset as described in **Table A 2** and **Table A 3**, respectively and listed in **Listing 3**.

Smoking history, medical history, prior and concomitant medication, exhaled carbon monoxide, drug/alcohol test, skin prick test and tobacco consumption will be listed by subject in **Listing 4** to **Listing 10**, respectively.

#### 5.5.3 Primary analysis

STT for each time point will be summarized by smoker and never smoker groups using the descriptive statistics: mean, median, standard deviation, quartiles (Q1 and Q3), minimum and maximum values and 95% confidence interval (CI).

Changes in STT from T0 will be computed at T4, T8 and T12 and summarized by smoker and never smoker group using the descriptive statistics: mean, minimum, maximum, median, quartiles (Q1 and Q3), standard deviation (SD) and 95% confidence interval (CI).

The plasma nicotine levels for each time point will be summarized by smoker and never smoker group using the descriptive statistics mean, minimum, maximum, median, quartiles, standard deviation (SD) and 95% confidence interval (CI). The relationship between plasma nicotine levels and STT at each time point will be evaluated by spearman correlation as well as graphical presentation of these endpoints by time point and smoker and never smoker group.

Results regarding STT, plasma nicotine and STT versus plasma nicotine will be presented for FAS and PP dataset as described in **Table A 4** to **Table A 8** and in **Figure A 1** to **Figure A 4**.

Data regarding STT test will be listed by subject in **Listing 11**.

#### 5.5.4 Secondary analysis

#### 5.5.4.1 Nasal scraping procedures

Descriptive statistics of RNA results will be summarized by smoker and never smoker groups using total number of observations (n), mean, median, standard deviation, quartiles (Q1 and Q3) and minimum and maximum values.

Nasal scraping procedures will be presented for FAS dataset as described in Table A 9.

#### 5.5.4.2 Safety analysis

Vital signs (systolic blood pressure, diastolic blood pressure, pulse rate and respiratory rate) will be summarized by total number of observations (n), mean, median, standard deviation, quartiles (Q1 and Q3) and minimum and maximum values.

An overall summary of AEs will be presented by smoker and never smoker groups showing the number of events and percent of study participants who experienced AEs, SAEs, severe AEs and AEs leading to study discontinuation.

A summary of AEs by System Organ Class (SOC) and Preferred Term (PT) according to Medical Dictionary for Regulatory Activities (MedDRA) by smoker and never smoker groups will be presented.

Each parameter of hematology, clinical chemistry and urine will be summarized over time by smoker and never smoker group thought total number of observations (n), mean, median, standard deviation, quartiles (Q1 and Q3) and minimum and maximum values. Number (n) and frequency distribution (%) of normal and abnormal values will also be present by each parameter.

All safety analyses will be performed for the safety dataset only.

Vital signs measures will be presented for safety dataset in Table A 10 and listed in Listing 12

Incidence and frequency distribution of AEs, SAEs, AEs with reasonable possibility of relationship with study drug will be presented in **Table A 11** and **Table A 12**. All adverse events and serious adverse events will also be listed by subject in **Listing 13** and **Listing 14**.

Regarding laboratory parameters, results of hematology, chemistry and urinalysis will be presented for safety dataset in **Table A 13**, **Table A 14** and **Table A 15** and listed by subject in **Listing 15**. Results on serology at visit 1 will be presented in **Table A 16**.

#### 5.6 Missing values

Missing STT values for a time point will be treated as missing. When STT detection takes longer than 1 hour, the STT will be considered as 1 hour. When the subject is not able to test saccharine on direct application, the STT values should be treated as missing, and these subjects should not be included in the STT analysis.

Regarding plasma nicotine samples:

- Missing sampling time: if the time of collection for a sample is unknown, that individual data point will be treated as missing data for descriptive statistics.
- Missing concentration data: missing concentration data will be treated as missing and replaced with a "." in the concentration dataset. No values will be imputed.
- Concentration data below lower limit of quantification (LLOQ=0.399 ng/mL): in the calculation
  of descriptive statistics for concentration data at each sampling time point, all LLOQ values will
  be treated as zero for time zero and as 1/2 LLOQ for the remaining time

#### 6 CLARIFICATIONS TO THE STUDY PROTOCOL

In the study protocol, the populations that should be considered in each statistical analysis is not clear. In this SAP the following assumptions were considered:

- Statistical analysis for demographics will be performed for the FAS and PP population;
- Primary analysis will be performed for the FAS and PP population;
- Safety analysis will be performed for the safety population.

#### 7 APPENDIX 1: DERIVED VARIABLES

The following variables will be derived:

Group of subjects – A dichotomous variable (smoker/never smoke) will be calculated.

Smoker – subjects who meet all of the following criteria at Visit 1 and at Visit 2:

- A positive urine cotinine test (=200 ng/mL).
- Smoked at least 20 cigarettes per day for at least the past 5 years.
- eCO levels >10 parts per million (ppm).
- No plans to quit smoking in the next 3 months.

Never smoker – subjects who meet all of the following criteria at Visit 1 and at Visit 2:

- Subject who has smoked less than 100 cigarettes throughout their lifetime and no cigarettes in the past 3 years.
- A negative urine cotinine test (<50 ng/mL).
- eCO levels = 5 ppm.

**STT** – At each time point, STT value will be obtained as the difference between end time and start time, in minutes, of STT test. When STT detection takes longer than 1 hour, the STT will be considered as 1 hour (60 minutes). When the subject is not able to test saccharine on direct application, the STT values should be treated as missing, and these subjects should not be included in the STT analysis.

#### 8 **APPENDIX 2: TABLES AND FIGURES**

#### Table A 1 - Subjects' disposition

| | Total | Smoker | Never smoker |
|---|---|---|---|
| No. of subjects included in the study, n (%) | | | |
| Subjects who completed the study, n (%) <sup>a</sup> Subjects who discontinued, n (%) <sup>a</sup> Adverse event Best interest for study participant Non-compliance with study procedures Study terminated by investigator Study terminated by sponsor Withdrawal by subject Other | | | |
| Analysis populations, n (%) <sup>a</sup> FAS PP Safety | | | |

FAS: Full analysis set. PP: Per protocol. a) Percentages calculated within included subjects.

Table A 2 – Demographic and anthropometric characteristics at visit 1 – FAS population

| Smoker<br>(n=xx) | Never smoker (n=xx) |
|------------------|---------------------|

# Age (years) N Mean

Median

Median Standard Deviation Q1 Q3 Minimum Maximum

# Gender, n (%) Male Female

Total

#### Ethnicity, n (%)

Hispanic or Latino

Not Hispanic or Latino

Total

#### Race, n (%)

American Indian or Alaska native

Black or African American Native Hawaiian / other pacific islander

Total

# Height (cm) N Mean

Median

Standard Deviation

Q1 Q3

Minimum

Maximum

### Weight (kg) N

Mean

Median

Standard Deviation

Q1 Q3 Minimum

Maximum

#### BMI (kg/m²)

Ν

Mean

Median

Standard Deviation

Minimum

Maximum

BMI: body mass index.

Table A 3 – Demographic and anthropometric characteristics at visit 1 – PP population

| | Smoker<br>(n=xx) | Never smoker (n=xx) |
|---|---|---|
| Age (years) | | |
| N | | |
| Mean | | |
| Median | | |
| Standard Deviation<br>Q1 | | |
| Q3 | | |
| Minimum | | |
| Maximum | | |
| Gender, n (%) Male Female Total | | |
| Ethnicity, n (%) Hispanic or Latino Not Hispanic or Latino Total | | |
| Race, n (%) Asian American Indian or Alaska native Black or African American Native Hawaiian / other pacific islander White | | |

# Height (cm) N Mean Median

Standard Deviation

Q1 Q3 Minimum Maximum

Weight (kg) N Mean Median Standard Deviation Q1 Q3 Minimum Maximum

#### BMI (kg/m²)

N Mean

Median

Standard Deviation

Q1 Q3 Minimum

Maximum

BMI: body mass index.

Table A 4 – Saccharin transit time – FAS population

| | Visit 1 | | V | isit 2 | Vis | it 3 –T0 | Visi | it 3 – T4 | Visit 3 – T8 | | Visit | 3 – T12 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Smoker<br>(n=xx) | Never<br>smoker<br>(n=xx) | Smoker<br>(n=xx) | Never<br>smoker<br>(n=xx) | Smoker<br>(n=xx) | Never<br>smoker<br>(n=xx) | Smoker<br>(n=xx) | Never<br>smoker<br>(n=xx) | Smoker<br>(n=xx) | Never<br>smoker<br>(n=xx) | Smoker<br>(n=xx) | Never<br>smoke<br>(n=xx) |
| TT result (min) N Mean Median Standard Deviation Q1 Q3 Minimum Maximum | | | | | | | | | | | | |
| 95% CI | | | | | | | | | | | | |
| hange from T0 | | | | | | | | | | | | |
| N | _ | _ | _ | _ | _ | _ | | | | | | |
| Mean | _ | - | - | _ | - | - | | | | | | |
| Median | _ | - | - | _ | - | - | | | | | | |
| Standard Deviation | _ | - | - | _ | - | - | | | | | | |
| Q1 | _ | _ | _ | _ | _ | _ | | | | | | |
| Q3 | _ | _ | _ | _ | _ | _ | | | | | | |
| ~~· | _ | _ | _ | _ | _ | _ | | | | | | |
| Minimum | | | | | | | | | | | | |

STT value will be obtained as the difference between end time and start time, in minutes (see appendix 1).

Table A 5 – Saccharin transit time – PP population

| | Visit 1 | | Visit 2 | | Vis | Visit 3 –T0 | | Visit 3 – T4 | | Visit 3 – T8 | | Visit 3 - T12 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Smoker<br>(n=xx) | Never<br>smoker<br>(n=xx) | Smoker<br>(n=xx) | Never<br>smoker<br>(n=xx) | Smoker<br>(n=xx) | Never<br>smoker<br>(n=xx) | Smoker<br>(n=xx) | Never<br>smoker<br>(n=xx) | Smoker<br>(n=xx) | Never<br>smoker<br>(n=xx) | Smoker<br>(n=xx) | Never<br>smoker<br>(n=xx) |
| STT result (min) N Mean Median Standard Deviation Q1 Q3 Minimum Maximum | | | | | | | | | | | | |
| 95% CI | | | | | | | | | | | | |
| Change from T0 | | | | | | | | | | | | |
| N | - | - | _ | _ | _ | _ | | | | | | |
| Mean | _ | _ | _ | _ | _ | _ | | | | | | |
| Median | _ | _ | _ | _ | _ | _ | | | | | | |
| Standard Deviation | _ | _ | _ | _ | _ | _ | | | | | | |
| Q1 | _ | _ | _ | _ | _ | _ | | | | | | |
| Q3 | _ | _ | _ | _ | _ | _ | | | | | | |
| Minimum | _ | _ | _ | _ | _ | _ | | | | | | |
| Maximum | - | - | - | - | - | - | | | | | | |
| 95% CI | | | | | | | | | | | | |

STT value will be obtained as the difference between end time and start time, in minutes (see appendix 1).

Table A 6 – Plasma nicotine sample at Visit 3 – FAS population

| | Visit 3 –T0 | | Visit 3 – T4 | | Visit 3 – T8 | | Visit 3 – T12 | 2 |
|---|---|---|---|---|---|---|---|---|
| | Smoker<br>(n=xx) | Never smoker (n=xx) | Smoker<br>(n=xx) | Never smoker (n=xx) | Smoker<br>(n=xx) | Never smoker (n=xx) | Smoker<br>(n=xx) | Never smoker (n=xx) |
| Result (%) N Mean Median Standard Deviation Q1 Q3 Minimum Maximum 95% CI | | | | | | | | |

Table A 7 – Plasma nicotine sample at Visit 3 – PP population

| | Visit 3 -T0 | | Visit 3 – T4 | | Visit 3 – T8 | | Visit 3 - T12 | |
|---|---|---|---|---|---|---|---|---|
| | Smoker<br>(n=xx) | Never smoker (n=xx) | Smoker<br>(n=xx) | Never smoker (n=xx) | Smoker<br>(n=xx) | Never smoker (n=xx) | Smoker<br>(n=xx) | Never smoker (n=xx) |
| Result (%) N Mean Median Standard Deviation Q1 Q3 Minimum Maximum | | | | | | | | |
| 95% CI | | | | | | | | |

#### Table A 8 - Plasma nicotine sample versus STT

| FAS | population | PP population | |
|---|---|---|---|
| Smoker<br>(n=xx) | Never smoker (n=xx) | Smoker<br>(n=xx) | Never smoker (n=xx) |

#### Plasma nicotine vs STT at Visit 3 - T0

p-value Spearman correlation coefficient

#### Plasma nicotine vs STT at Visit 3 - T4

p-value Spearman correlation coefficient

#### Plasma nicotine vs STT at Visit 3 - T8

p-value Spearman correlation coefficient

#### Plasma nicotine vs STT at Visit 3 - T12

p-value Spearman correlation coefficient

STT: Saccharin transit time.



Figure A 1 – Plasma nicotine levels versus STT by smokers and never smokers, at T0 – FAS population



Figure A 2 – Plasma nicotine levels versus STT by smokers and never smokers, at T4 – FAS population



Figure A 3 – Plasma nicotine levels versus STT by smokers and never smokers, at T8 – FAS population



Figure A 4 – Plasma nicotine levels versus STT by smokers and never smokers, at T12 – FAS population

#### Table A 9 - Nasal scraping at visit 3 - FAS population

| Total<br>(n=xx) |
|-----------------|

Method, n (%) Left nostril (method 1) Right nostril (method 2) Total

# Only method 1 (5 subjects) RNA N

Mean

Median

Standard Deviation

Q1 Q3 Minimum

Maximum

### Only method 2 (5 subjects)

N Mean

Median

Standard Deviation

Q1 Q3 Minimum Maximum

#### Method 1 or 2 (10 subjects)

#### RNA

Mean

Median

Standard Deviation

Q1 Q3 Minimum Maximum

#### Method 1 and 2 (4 subjects)

#### RNA

Mean Median Standard Deviation

Q1 Q3

Minimum Maximum

#### Table A 10 - Vital signs - Safety population

| Visit 1 | | Visit 2 | | Visit 3 | |
|---|---|---|---|---|---|
| Smoker<br>(n=xx) | Never<br>smoker<br>(n=xx) | Smoker<br>(n=xx) | Never<br>smoker<br>(n=xx) | Smoker<br>(n=xx) | Never<br>smoker<br>(n=xx) |

#### Systolic blood pressure (mmHg)

N Mean Median

Standard Deviation

Q1 Q3

Minimum Maximum

#### Diastolic blood pressure (mmHg)

N Mean

Median

Standard Deviation

Q1 Q3

Minimum Maximum

#### Pulse rate (beats/min)

N Mean

Mean Median Standard Deviation Q1 Q3 Minimum Maximum

#### Respiratory rate (breaths/min)

N Mean Median Standard Deviation

Q1 Q3 Minimum

Maximum

#### Table A 11 – Overall summary of adverse events – Safety population

| Smoker<br>(n=xx) | | Never smoker<br>(n=xx) | |
|------------------|------|------------------------|------|
| n (%) | nAEs | n (%) | nAEs |

Any adverse event, n (%)
Any serious adverse event, n (%)
Any severe adverse event, n (%)
Any adverse event leading to study discontinuation, n (%)

n (%) = Number (percent) of subjects. nAE = Number of adverse events.

#### Table A 12 - Adverse events - Safety population

| Smoker<br>(n=xx) | | Never sm<br>(n=xx) | oker |
|------------------|--------|--------------------|---------------|
| n (%) | nAEs | n (%) | nAEs |
| | (n=xx) | (n=xx) | (n=xx) (n=xx) |

n (%) = Number (percent) of subjects. nAE = Number of adverse events.

#### Table A 13 – Hematology – Safety population

| Visit 1 | | Visit 3 | |
|---|---|---|---|
| Smoker<br>(n=xx) | Never smoker (n=xx) | Smoker<br>(n=xx) | Never smoker (n=xx) |

#### Hematocrit (unit)

Mean

Median

Standard Deviation

Q1 Q3

Minimum

Maximum

#### Normal/abnormal, n (%)

Normal

Abnormal

Total

#### Hemoglobin (unit)

Mean

Median

Standard Deviation

Q1

Q3 Minimum

Maximum

#### Normal/abnormal, n (%)

Normal Abnormal Total

#### MCH (unit)

Mean

Median Standard Deviation

Q1 Q3

Minimum

Maximum

#### Normal/abnormal, n (%)

Normal

Abnormal

Total

#### MCHC (unit)

Mean

Median

Standard Deviation

Q3

Minimum

Maximum

#### Normal/abnormal, n (%)

Normal

Abnormal Total

#### MCV (unit)

Mean

Median Standard Deviation

Q1

Q3

Minimum

Maximum

#### Normal/abnormal, n (%)

Normal

**Abnormal** 

Total

#### Platelet count (unit)

Mean

Median

Standard Deviation

Q1

Q3

Minimum

Maximum

#### Normal/abnormal, n (%)

Normal

Abnormal

Total

#### RBC (unit)

Mean

Median

Standard Deviation

Q1 Q3

Minimum

Maximum

#### Normal/abnormal, n (%)

Normal

Abnormal Total

#### WBC (unit)

Mean Median Standard Deviation

Q1

Q3

Minimum

Maximum

#### Normal/abnormal, n (%)

Normal

Abnormal

Total

#### Neutrophils (unit)

Mean

Median

Standard Deviation

Q1

Q3

Minimum

Maximum

#### Normal/abnormal, n (%)

Normal

Abnormal

Total

#### Basophils (unit)

N Mean Median

Standard Deviation

Q1 Q3

Minimum Maximum

#### Normal/abnormal, n (%)

Normal

Abnormal

Total

#### **Eosinophils (unit)**

Mean

Median

Standard Deviation Q1 Q3 Minimum Maximum

#### Normal/abnormal, n (%)

Normal Abnormal Total

# Lymphocytes (unit) N Mean

Median Standard Deviation

Q1 Q3

Minimum Maximum

# Normal/abnormal, n (%) Normal Abnormal

Total

#### Monocytes (unit)

N Mean

Mean Median Standard Deviation Q1 Q3 Minimum Maximum

# Normal/abnormal, n (%) Normal Abnormal Total

#### Table A 14 - Clinical chemistry - Safety population

| | Visit 1 | | Visit 3 |
|---|---|---|---|
| Smoker<br>(n=xx) | Never smoker (n=xx) | Smoker<br>(n=xx) | Never smoker<br>(n=xx) |

#### Albumin (unit)

N Mean

Median

Standard Deviation

Q1 Q3

Minimum

Maximum

#### Normal/abnormal, n (%)

Normal Abnormal Total

#### Total protein (unit)

Mean

Median

Standard Deviation

Q1

Q3 Minimum

Maximum

#### Normal/abnormal, n (%)

Normal Abnormal Total

#### AP (unit)

Mean

Median

Standard Deviation

Q1 Q3

Minimum

Maximum

#### Normal/abnormal, n (%)

Normal

Abnormal

Total

#### ALT (unit)

Mean

Median

Standard Deviation

Q1

Q3

Minimum

Maximum

#### Normal/abnormal, n (%)

Normal

Abnormal Total

#### AST (unit)

Mean Median Standard Deviation

Q1

Q3

Minimum

Maximum

#### Normal/abnormal, n (%)

Normal

**Abnormal** 

Total

#### BUN (unit)

Mean

Median

Standard Deviation

Q1

Q3

Minimum

Maximum

#### Normal/abnormal, n (%)

Normal

Abnormal

Total

#### Creatinine (unit)

Mean

Median

Standard Deviation

Q1 Q3

Minimum

Maximum

#### Normal/abnormal, n (%)

Normal

Abnormal Total

#### Fasting glucose (unit)

Mean Median Standard Deviation

Q1

Q3

Minimum

Maximum

#### Normal/abnormal, n (%)

Normal

Abnormal

Total

#### Fibrinogen (unit)

Mean

Median

Standard Deviation

Q1

Q3

Minimum

Maximum

#### Normal/abnormal, n (%)

Normal

Abnormal

Total

#### GGT (unit)

Ν

Mean

Median Standard Deviation

Q1 Q3 Minimum

Maximum

#### Normal/abnormal, n (%)

Normal

Abnormal

Total

#### LDH (unit)

Mean

Median
Standard Deviation

Q1 Q3 Minimum

Maximum

### Normal/abnormal, n (%)

Normal

Abnormal

Total

### Potassium (unit)

Mean

Median

Standard Deviation

Q1 Q3

Minimum

Maximum

### Normal/abnormal, n (%)

Normal

Abnormal

Total

### Sodium (unit)

Mean

Median

Standard Deviation

Q1 Q3 Minimum

Maximum

### Normal/abnormal, n (%) Normal

Abnormal

Total

### Total bilirubin (unit)

Mean

Median

Standard Deviation

Q3

Minimum

Maximum

### Normal/abnormal, n (%)

Normal

Abnormal

Total

### Direct bilirubin (unit)

Mean

Median

Standard Deviation

Q1 Q3

Minimum

Maximum

### Normal/abnormal, n (%)

Normal Abnormal

Total

### Total cholesterol (unit)

Mean

Median

Standard Deviation

Q1 Q3

Minimum

Maximum

Normal/abnormal, n (%) Normal Abnormal Total

### Triglycerides (unit)

N
Mean
Median
Standard Deviation
Q1
Q3
Minimum
Maximum Maximum

### Normal/abnormal, n (%) Normal

Abnormal Total

AP: Alkaline phosphatase. ALT: alanine aminotransferase. AST: aspartate aminotransferase. BUN: blood urea nitrogen. GGT: Gamma-glutamyl transferase. LDH: lactate dehydrogenase.

### Table A 15 – Urine – Safety population

| V | isit 1 | | Visit 3 |
|---|---|---|---|
| Smoker<br>(n=xx) | Never smoker (n=xx) | Smoker<br>(n=xx) | Never smoker (n=xx) |

рΗ

Mean Median

Standard Deviation

Q1 Q3

Minimum Maximum

### Normal/abnormal, n (%)

Normal Abnormal

### Bilirubin (unit)

Mean

Total

Median

Standard Deviation

Q1

Q3 Minimum

Maximum

## Normal/abnormal, n (%) Normal Abnormal Total

### Glucose (unit)

Mean

Median Standard Deviation

Q1 Q3

Minimum

Maximum

### Normal/abnormal, n (%)

Normal

Abnormal

Total

### Nitrite (unit)

Mean

Median

Standard Deviation

Q1

Q3

Minimum Maximum

### Normal/abnormal, n (%)

Normal

Abnormal Total

### Red blood cells trace (unit)

N Mean Median Standard Deviation

Q1

Q3

Minimum

Maximum

### Normal/abnormal, n (%)

Normal

**Abnormal** 

Total

### Protein (unit)

N Mean Median Standard Deviation

Q1 Q3 Minimum Maximum

## Normal/abnormal, n (%) Normal Abnormal Total

### Specific gravity (unit)

N Mean Median Standard Deviation

Q1 Q3 Minimum Maximum

# Normal/abnormal, n (%) Normal Abnormal Total

### Table A 16 – Serology at visit 1 – Safety population

| | Smoker<br>(n=xx) | Never smoker<br>(n=xx) |
|---|---|---|
| Hepatitis B surface antigen, n (%) | | |
| Positive | | |
| Negative | | |
| Total | | |
| Hepatitis C virus, n (%) | | |
| Positive | | |
| Negative | | |
| Total | | |
| Anti-HIV1/2, n (%) | | |
| Positive | | |
| Negative | | |
| Total | | |

HIV: human immunodeficiency virus.

### 9 APPENDIX 2: LISTINGS

### Listing 1 – Subjects' disposition

| Subject Subject complete the Reason for study discontinuation | Group | FAS | PP | Safety |
|---|---|---|---|---|
|---|---|---|---|---|

### Listing 2 – Protocol deviations

| Subject Protocol deviation | Group | FAS | PP | Safety |
|----------------------------|-------|-----|----|--------|
|----------------------------|-------|-----|----|--------|

### Listing 3 – Demographic and anthropometric characteristics at visit 1

| Subject | Age | Sex | Ethnicity | Race | Height (cm) | Weight (kg) | BMI (kg/m²) | Group | FAS | PP | Safety |
|---|---|---|---|---|---|---|---|---|---|---|---|

### Listing 4 – Smoking history

| Subject 100 cigarettes or to qu | Subject smoked at least 20 cigarettes per day for at least the past 5 consecutive years | No. of years<br>that subject<br>smoked<br>cigarettes in<br>their entire life | No. of<br>cigarettes<br>smoked<br>per day | Subject mostly<br>exhales smoke<br>through the<br>nose | Use of E-<br>cigarette over<br>the last 3<br>months | Use of Cigar<br>over the last 3<br>months | Use of Pipe or<br>hookah over<br>the last 3<br>months |
|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|

| Use of Snuff or<br>Chewing Tobacco<br>over the last 3 months | Use of Nicotine product to help quit smoking over the last 3 months | Use of other over the last 3 months | Use of other tobacco/nicotine containing products over the last 3 months | Subject smoked any cigarettes or more in the past 3 years | Use of E-<br>cigarette over<br>the last 3 years | Use of Cigar<br>over the last 3<br>years | Use of Pipe or<br>hookah over<br>the last 3<br>years |
|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|

| Use of Snuff or<br>Chewing Tobacco<br>over the last 3 years | Use of Nicotine product to help quit smoking over the last 3 years | Use of other over the last 3 years | Use of other tobacco/nicotine containing products over the last 3 years | Brand of cigarettes | Group | FAS | PP | Safety |
|---|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|---|

### Listing 5 – Medical history

| Subject | MH<br>subcategory | MH term | Start date | Ongoing | End date | Group | FAS | PP | Safety |
|---|---|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|---|---|

### Listing 6 – Prior and concomitant medication

| Subject | Medication | Dose | Dose<br>units | Frequency | Route | Start<br>date | ongoing | End<br>date | Indication | Used to<br>treat AE or<br>MH? | AE or<br>MH | Group | FAS | PP | Safety |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|

AE: Adverse event. MH: Medical history. FAS: Full analysis set. PP: Per protocol.

### Listing 7 – Exhaled Carbon Monoxide

| Carbott Visit Confection date Extracted Carbott Monoxide lever (ppm) | Subject | Visit | Collection date | Exhaled Carbon Monoxide level (ppm) | Group | FAS | PP | Safety |
|---|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|---|

### Listing 8 - Drug/alcohol test

| Subject Collection time Panel name Test name Result Group FAS PP Safe | Subject | ame Test name | Result Group | FAS | PP | Safety |
|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|

### Listing 9 - Skin prick test

| Subject | Skin prick test<br>date | Allergen | Mean wheal<br>diameter (mm) | Group | FAS | PP | Safety |
|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|

### Listing 10 – Tobacco consumption

| Subject | Visit | Current use of tobacco | Tobacco consumption date | Tobacco consumption time | Group | FAS | PP | Safety |
|---|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|---|

### Listing 11 – Saccharin transit time test

| Subject | Visit | Date | STT test performed | STT test date | Start<br>time | End<br>time | Was the subject able to perceive sweet taste within 60 minutes time? | Did the study participant taste the saccharin after direct application? | Group | FAS | PP | Safety |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|---|---|---|---|---|

STT: Saccharin transit time. FAS: Full analysis set. PP: Per protocol.

### Listing 12 – Vital signs

| Subject | Visit | Systolic blood pressure (mmHg) | Diastolic blood pressure (mmHg) | Pulse rate (beats/min) | Respiratory rate (breaths/min) | Group | FAS | PP | Safety |
|---|---|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|---|---|

### Listing 13 – Adverse events

| Subject | AE | Start<br>date | ongoing | End<br>date | Serious | Severity | Relationship to study procedures | Action taken | Outcome | Study<br>discontinuation | Group | FAS | PP | Safety |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|

AE: Adverse event. FAS: Full analysis set. PP: Per protocol.

### Listing 14 - Serious adverse events

| Subject | AE | Congenital anomaly or birth defect | Significant<br>disability | Death | Hospitalization | Life<br>threatening | Other medical important event | Group | FAS | PP | Safety |
|---|---|---|---|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|---|---|---|---|

AE: Adverse event. FAS: Full analysis set. PP: Per protocol.

### Listing 15 – Labs (hematology, chemistry and urine analysis)

| Subject | Collection date | Panel<br>name | Test name | Result | Normal<br>range | Normal<br>range<br>indicator | Clinically significant | Is abnormal test result related with an adverse event or concomitant medication? | Group | FAS | PP | Safety |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|---|---|---|---|---|